CLINICAL TRIAL: NCT01701882
Title: A Pilot Study to Assess the Feasibility of Switching, Individuals Receiving Atripla With Continuing Central Nervous System (CNS) Toxicity, to a Fixed Dose Combination of Tenofovir/Emtricitabine/Rilpivirine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSAT 047
Record Dates: First submitted 2012-09-19; First posted 2012-10-05 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: HIV
MeSH Terms: interventions — Tenofovir

ARMS (1):
- tenofovir/emtricitabine/rilpivirine (Experimental): A one pill fixed dose combination of tenofovir 245mg, emtricitabine 200mg and rilpivirine 25mg once daily.
  Interventions: Drug: tenofovir/emtricitabine/rilpivirine

INTERVENTIONS:
Drug: tenofovir/emtricitabine/rilpivirine

SUMMARY:
The purpose of the study is to investigate the benefits of switching away from efavirenz (which patients are taking in combination with Kivexa® or as part of the combination pill, Atripla®) in patients with central nervous system side effects (such as insomnia {difficulty with sleeping}, bad dreams etc). The investigators in this study will investigate the effect of switching to a single tablet regimen (Eviplera®) containing tenofovir, emtricitabine and rilpivirine. If patients are currently taking Atripla, rilpivirine will be the only new component of the combination.

Rilpivirine is a drug for HIV treatment, licensed for first-line treatment. In combination with Truvada®, it showed fewer side effects when compared to efavirenz in 2 other clinical studies, where patients were starting HIV treatment for the first time.

This study will also investigate the safety (in terms of other side effects and the routine blood tests which we ordinarily use to monitor your treatment) and monitor effectiveness, your viral load and CD4 counts, when you switch treatment to tenofovir/emtricitabine/rilpivirine.

ELIGIBILITY:
Inclusion Criteria:

* Patient volunteers who meet all of the following criteria are eligible for this trial:

  1. Is male or female aged 18 years or above
  2. Has HIV-1 infection documented in their medical notes
  3. Has signed the Informed Consent Form voluntarily
  4. Is willing to comply with the protocol requirements
  5. Has been on Atripla for at least 12 weeks OR Kivexa plus efavirenz
  6. Has an HIV-plasma viral load at screening <50 copies/mL (single re-test allowed)
  7. Has a CD4 cell count at screening >50 cells/mm3
  8. Estimated glomerular filtration rate (MDRD) >50 ml/min.
  9. Has symptomatic CNS related toxicity associated with EFV
  10. If female and of childbearing potential, is using effective birth control methods (as agreed by the investigator) and is willing to continue practising these birth control methods during the trial and for at least 30 days after the end of the trial. Note: Women who are postmenopausal for least 2 years, women with total hysterectomy, and women who have a tubal ligation are considered of non-childbearing potential
  11. If a heterosexually active male, he is using effective birth control methods and is willing to continue practising these birth control methods during the trial and until follow-up visit

      Exclusion Criteria:
* Patients meeting 1 or more of the following criteria cannot be selected:

  1. Infected with HIV-2
  2. Using any concomitant therapy disallowed as per SPC for the study drugs (note acid-reducing agents and interaction with rilpivirine)
  3. Has acute viral hepatitis including, but not limited to, A, B, or C
  4. Has chronic hepatitis B and/or C with AST and/or ALT >5 x ULN Note: Subjects can enter trial with chronic HBV if HBV-DNA undetectable at screen (and no detectable result in last 6 months) and with chronic HCV if not expected to require treatment during the trial period.
  5. Any investigational drug within 30 days prior to the trial drug administration
  6. Has received rilpivirine in the past
  7. Any clinical evidence of baseline resistance mutations
  8. Known allergy to lactose monohydrate, sunset yellow aluminium lake (E110), and patients with galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption
  9. Severe hepatic impairment
  10. Moderate or severe renal impairment (creatinine clearance < 50ml/min)
  11. If female, she is pregnant or breastfeeding
  12. Screening blood result with any grade 3/4 toxicity according to Division of AIDS (DAIDS) grading scale, except: asymptomatic grade 3 glucose, amylase or lipid elevation or asymptomatic grade 4 triglyceride elevation (re-test allowed).
  13. Any condition (including drug/alcohol abuse) or laboratory results which, in the investigator's opinion, interfere with assessments or completion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Resolution of toxicity after 12 weeks | 12 weeks
  To investigate whether switching individuals with intolerance to efavirenz-containing cART (as Atripla or Kivexa plus Efavarinz) to tenofovir/emtricitabine/rilpivirine is associated with resolution of toxicity after 12 weeks. CNS toxicity will be measured by a questionnaire based on efavirenz SPC and graded based on the ACTG adverse event scale.

SECONDARY OUTCOMES:
Resolution of toxicity after 24 weeks | 24 weeks
  To investigate whether switching to tenofovir/emtricitabine/rilpivirine is associated with resolution of toxicity after 24 weeks. CNS toxicity will be measured by a questionnaire based on efavirenz SPC and graded based on the ACTG adverse event scale.

CONTACTS AND LOCATIONS:
Locations (1):
- St Stephen's AIDS Trust, London, United Kingdom